CLINICAL TRIAL: NCT04355377
Title: Hepatic Artery From Origin to Segmental Branching: a 500 Case CT Study
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PI250
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-04

CONDITIONS: Hepatic Artery
Keywords: Hepatic Artery; Anatomy; MDCT

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients
  Interventions: Other: Non intervention

INTERVENTIONS:
Other: Non intervention — Non intervention

SUMMARY:
The origin of the hepatic artery is known to be highly variable, as reported by Michels in 1966 and other authors. This variability has an indisputable impact regarding hepatic, pancreatic and upper gastro-intestinal surgery.

As the investigators go deeper into the liver's parenchyma, full-liver and segment IV studies have also found high levels of variability. Only few cadaveric studies have analyzed the entire liver and with limited sample size.

The current CT technology allows for an accurate analysis of the arterial branching thanks to the 0.625mm voxel.

The aim of this CT study is to describe the anatomy of hepatic arterial segmental branching from the origin of the hepatic artery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing CT with arterial abdominal imaging

Exclusion Criteria:

* imaging with radiological artefact (movement, biliary prothesis,..)
* hepatic resection (except small non anatomic resections)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Systematic inclusion of patients undergoing CT imaging with arterial abdominal contrast between November 2019 and April 2020
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Anatomic description of the hepatic artery | November 1rst 2019 to May, 30 2020
  Analysis of 0.625mm voxel CT

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No